CLINICAL TRIAL: NCT01824290
Title: A Double-Blind Efficacy and Safety Study of the Phosphodiesterase Type 5 Inhibitor Tadalafil in Pediatric Patients With Pulmonary Arterial Hypertension
Brief Title: A Study of Tadalafil in Pediatric Participants With Pulmonary Arterial Hypertension (PAH)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 10609; H6D-MC-LVHV (Other: Eli Lilly and Company); 2012-002354-23 (EudraCT Number)
Record Dates: First submitted 2013-04-01; First posted 2013-04-04 (Estimated); Results first posted 2020-03-23 (Actual); Last update posted 2021-11-05 (Actual); Status verified 2021-11

CONDITIONS: Hypertension, Pulmonary
MeSH Terms: conditions — Hypertension, Pulmonary | interventions — Tadalafil

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Tadalafil (Experimental): Period 1: 20 mg or 40 mg administered orally by tablets once a day.
  Period 2: 20 mg for middle weight and 40 mg for heavy weight administered orally by tablets once a day.
  Final tadalafil doses for Period 1 (6-month double-blind) were assigned after the weight cohort completion from H6D-MC-LVIG (NCT01484431).Tadalafil doses would range from 5 milligram (mg) to 40 mg depending on body weight cohorts. Heavy weight cohort ≥40 kilogram (kg), Middle weight cohort ≥25 kg to <40 kg: administered orally by tablets once a day. Light weight cohort <25 kg: administered orally by suspension once a day.
  Participants receiving tadalafil in Period 1 continued to receive tadalafil during Period 2 (2-year open-label extension).
  Interventions: Drug: Tadalafil; Drug: ERA as specific PAH treatment
- Placebo (Placebo Comparator): Period 1: Participants received placebo orally by tablets once a day.
  Period 2: 20 mg for middle weight and 40 mg for heavy weight administered orally by tablets once a day.
  Final placebo dose for Period 1 (6-month double-blind) was be assigned after the weight cohort completion from H6D-MC-LVIG (NCT01484431) to maintain blinding depending on body weight cohort.
  Participants receiving placebo in Period 1 Period 2 (2-year open-label extension) would receive tadalafil in Period 2 at the corresponding tadalafil dose in that participant's weight group.
  Interventions: Drug: Placebo; Drug: ERA as specific PAH treatment

INTERVENTIONS:
Drug: Tadalafil — Administered orally by tablet form for heavy and middle weight participants. Administered orally by suspension for light weight participants.
  Other Names: LY450190; Cialis; Adcirca; IC351
  Arms: Tadalafil
Drug: Placebo — Administered orally by tablet for heavy and middle weight participants. Administered orally by suspension for light weight participants.
  Arms: Placebo
Drug: ERA as specific PAH treatment — All participants were taking endothelin receptor antagonist (ERA) (such as bosentan, ambrisentan and macitentan).

SUMMARY:
The main purpose of this study is to evaluate the safety and efficacy of tadalafil in pediatric participants with pulmonary arterial hypertension. Participants will receive study treatment for 6 months in the double-blind period (Period 1), and then will be eligible to enroll into an open-label 2 year extension period (Period 2) during which participants will receive tadalafil.

ELIGIBILITY:
Inclusion Criteria:

* ≥6 months to <18 years of age at screening
* Currently have a diagnosis of PAH that is either:

  * idiopathic, including hereditary
  * related to connective tissue disease
  * related to anorexigen use
  * associated with surgical repair of at least 6-month duration of congenital systemic to pulmonary shunt (eg, atrial septal defect, ventricular septal defect, patent ductus arteriosus)
* Have a history of a diagnosis of PAH established by a resting mean pulmonary artery pressure (mPAP) ≥25 millimeter of mercury (mm Hg), pulmonary artery wedge pressure ≤15 mm Hg, and a pulmonary vascular resistance (PVR) ≥3 Wood units via right heart catheterization (RHC). In the event that a pulmonary artery wedge pressure cannot be obtained during RHC, participants with a left ventricular end diastolic pressure (LVEDP) <15 mm Hg, with normal left heart function, and absence of mitral stenosis on echocardiography can be eligible for enrollment
* Have a World Health Organization (WHO) functional class value of II or III at the time of screening
* All participants must be receiving an endothelin receptor antagonist (ERA) (such as bosentan or ambrisentan) and must be on a maintenance dose with no change in dose (other than weight-based adjustments) for at least 12 weeks prior to screening and have a screening aspartate transaminase (AST)/alanine transaminase (ALT) <3 times the upper limit of normal (ULN)
* If on conventional PAH medication, including but not restricted to, anticoagulants, diuretics, digoxin, and oxygen therapy, the participant must be on stable doses with no changes (other than weight-based adjustments) for at least 4 weeks before screening
* Female participants of childbearing potential must test negative for pregnancy during screening. Furthermore, female participants must agree to abstain from sexual activity or to use two different reliable methods of birth control as determined by the Investigator during the study. Examples of reliable birth control methods include true abstinence as a lifestyle choice (periodic sexual abstinence method is not acceptable); the use of oral contraceptives; a reliable barrier method of birth control (diaphragms with contraceptive jelly; cervical caps with contraceptive jelly; condoms with contraceptive foam; intrauterine devices)
* Written informed consent from parents (and written assent from appropriately aged participants) will be obtained prior to any study procedure being performed

Exclusion Criteria:

* Have pulmonary hypertension related to conditions other than specified above, including but not limited to chronic thromboembolic disease, portal pulmonary hypertension, left-sided heart disease or lung disease and hypoxia
* History of left-sided heart disease, including any of the following:

  * clinically significant [pulmonary artery occlusion pressure (PAOP) 15-18 mm Hg] aortic or mitral valve disease (ie, aortic stenosis, aortic insufficiency, mitral stenosis, moderate or greater mitral regurgitation)
  * pericardial constriction
  * restrictive or congestive cardiomyopathy
  * left ventricular ejection fraction <40% by multigated radionucleotide angiogram (MUGA), angiography, or echocardiography
  * left ventricular shortening fraction <22% by echocardiography
  * life-threatening cardiac arrhythmias
  * symptomatic coronary artery disease within 5 years of study entry
* Unrepaired congenital heart disease
* Have a history of angina pectoris or other condition that was treated with long- or short-acting nitrates within 12 weeks before administration of study drug
* Have severe hepatic impairment, Child-Pugh Grade C
* Have severe renal insufficiency, defined as receiving renal dialysis or having a measured or estimated creatinine clearance (CC) <30 millimeter per minute (mL/min) (Schwartz Formula)
* Diagnosed with a retinal disorder (eg, hereditary retinal disorders, retinopathy of the preterm participant and other retinal disorders)
* Have severe hypotension or uncontrolled hypertension as determined by the Investigator
* Have significant parenchymal lung disease
* Have bronchopulmonary dysplasia
* Concurrent phosphodiesterase type 5 (PDE5) inhibitor therapy (sildenafil or vardenafil) or has received PDE5 inhibitor therapy within 12 weeks prior to the first study drug dosing
* Concurrent therapy with prostacyclin or its analogues within 12 weeks of screening
* Commenced or discontinued a chronic conventional PAH medication including but not restricted to: diuretics, anti-coagulants, digoxin, and oxygen therapy within 4 weeks of screening
* Currently receiving treatment with doxazosin, nitrates, or cancer therapy
* Current treatment with potent Cytochrome P450 3A4 (CYP3A4) inhibitors, such as antiretroviral therapy (protease inhibitor), systemic ketoconazole, or systemic itraconazole, or chronic use of potent CYP3A4 inducers, such as rifampicin
* Are nursing or pregnant
* Have previously completed or withdrawn from this study (LVHV), or any other study investigating tadalafil
* Have received tadalafil therapy within 12 weeks prior to the first study drug dosing or are hypersensitive to tadalafil
* Have allergy to the excipients, notably lactose
* Are currently enrolled in, or discontinued within the last 30 days from, a clinical trial involving an investigational product or non-approved use of a drug or device, or concurrently enrolled in any other type of medical research judged not to be scientifically or medically compatible with this study by the Sponsor
* Unable to take orally administered tablets (without chewing, crushing or breaking) or suspension
* Are Investigator site personnel directly affiliated with this study or their immediate families. Immediate family is defined as a spouse, parent, child or sibling, whether biological or legally adopted
* Diagnosis of Down syndrome

Ages: 6 Months to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 35 (Actual)
Dates: Start 2014-02-05 (Actual); Primary Completion 2019-03-18 (Actual); Study Completion 2021-03-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (43):
- United States (7):
  - Children's Heathcare of Atlanta, Inc. at Egleston, Atlanta, Georgia
  - Childrens Hospital of Michigan, Detroit, Michigan
  - Cincinnati Childrens Hospital Medical Center, Cincinnati, Ohio
  - Nationwide Children's Hosp, Columbus, Ohio
  - Vanderbilt Univeristy School of Medicine, Nashville, Tennessee
  - Texas Childrens Hospital, Houston, Texas
  - Primary Childrens Medical Center, Salt Lake City, Utah
- AKH, Vienna, Austria
- Universitaire Ziekenhuizen Leuven - Campus Gasthuisberg, Leuven, Belgium
- Brazil (4):
  - Pronto Socorro Cardiologico de Pernambuco-PROCAPE, Recife, Pernambuco
  - Irmandade da Santa Casa de Misericordia de Porto Alegre, Porto Alegre, Rio Grande do Sul
  - Instituto Dante Pazzanese de Cardiologia, São Paulo, São Paulo
  - UNIFESP - Escola Paulista de Medicina, São Paulo, São Paulo
- France (4):
  - CHU Hopital d'enfants de la Timone, Marseille
  - GH Necker - Enfants Malades, Paris
  - Hopital Haut Leveque - Group hospitalier Sud, Pessac
  - Chu de Toulouse - Hopital des Enfants, Toulouse
- Germany (2):
  - Universitätsklinikum Heidelberg, Heidelberg, Baden-Wurttemberg
  - Universitätsklinikum Ulm, Ulm, Baden-Wurttemberg
- Israel (2):
  - Sheba Medical Center, Tel Litwinsky, Ramat Gan
  - Schneider Medical Center, Petah Tikva
- Italy (3):
  - Istituto Giannina Gaslini Ospedale Pediatrico I.R.C.C.S., Genova, GE
  - Ospedale V. Monaldi, Napoli
  - Ospedale Bambino Gesu, Roma
- Japan (8):
  - Gunma Children's Medical Center, Shibukawa, Gunma
  - Asahikawa Medical College Hospital, Asahikawa, Hokkaido
  - Mie University Hospital, Tsu, Mie-ken
  - Okinawa Prefectural Nanbu Medical Center & Children's Med Ct, Haebaru-cho, Shimajiri-gun, Okinawa
  - Tokyo Metropolitan Children's Medical Center, Fuchū, Tokyo
  - Toho University Omori Medical Center, Ohta-Ku, Tokyo
  - National Center For Child Health And Development, Setagaya-ku, Tokyo
  - Shizuoka Prefectural Children's Hospital, Shizuoka
- Instituto Nacional de Cardiologia Ignacio Chavez, Mexico City, Mexico City, Mexico
- Universitair Medisch Centrum Groningen, Groningen, Netherlands
- Poland (4):
  - Instytut Pomnik-Centrum Zdrowia Dziecka, Warsaw, Woj Mazowieckie
  - Uniwersyteckie Centrum Kliniczne, Gdansk
  - Uniwersytecki Szpital Dzieciecy w Krakowie-Prokocimiu, Krakow
  - Wojewódzki Szpital Specjalistyczny we Wrocławiu, Wroclaw
- Spain (3):
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Hospital Universitario Ramon y Cajal, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
- Turkey (Türkiye) (2):
  - Hacettepe University Faculty of Medicine, Ankara
  - Gazi University Medical Faculty, Besevler/Ankara

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and EU, whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: https://vivli.org/

REFERENCES:
- See also: A Study of Tadalafil in Pediatric Participants With Pulmonary Arterial Hypertension (PAH) — https://trials.lillytrialguide.com/en-US/trial/5ejOJO01mwK2euskWAUoeu

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Per protocol and statistical analysis plan (SAP), the primary and secondary analysis from period 1 were performed to compare all tadalafil participants together versus all placebo participants together.
Groups:
- Placebo: Period 1: Participants received placebo orally by tablets once a day.
- Tadalafil: Period 1: 20 mg middle weight cohort or 40 mg for heavy weight cohort administered tadalafil orally by tablets once a day.
- Placebo/Tadalafil: Period 2: 20 mg middle weight cohort or 40 mg for heavy weight cohort administered tadalafil orally by tablets once a day.
  Participants had received placebo during period 1.
- Tadalafil/Tadalafil: Period 2: 20 mg middle weight cohort or 40 mg for heavy weight cohort administered tadalafil orally by tablets once a day.
  Participants had received tadalafil during period 1.
Period: Period 1: Double Blind
Arm/Group | Placebo | Tadalafil | Placebo/Tadalafil | Tadalafil/Tadalafil
Started | 18 | 17 | 0 | 0
Received at Least One Dose of Study Drug | 18 | 17 | 0 | 0
Received 20 mg | 0 | 4 | 0 | 0
Received 40 mg | 0 | 13 | 0 | 0
Completed | 15 | 15 | 0 | 0
Not Completed | 3 | 2 | 0 | 0
Not completed — Entry Criteria Not Met | 1 | 0 | 0 | 0
Not completed — Parent/Caregiver Decision | 1 | 1 | 0 | 0
Not completed — Investigator Reported Clinical Worsening | 1 | 1 | 0 | 0
Period: Period 2: Open-Label Treatment
Arm/Group | Placebo | Tadalafil | Placebo/Tadalafil | Tadalafil/Tadalafil
Started | 0 | 0 | 16 (As per the protocol, period 2 eligibility were participants who completed period 1 or experienced clinical worsening (CW) in period 1. 1 participant that had CW in period 1 continued to period 2.) | 16 (As per the protocol, period 2 eligibility were participants who completed period 1 or experienced clinical worsening (CW) in period 1. 1 participant that had CW in period 1 continued to period 2.)
Received 20 mg | 0 | 0 | 3 | 3
Received 40 mg | 0 | 0 | 13 | 13
Completed | 0 | 0 | 13 | 13
Not Completed | 0 | 0 | 3 | 3
Not completed — Adverse Event | 0 | 0 | 0 | 1
Not completed — Parent/caregiver Decision | 0 | 0 | 1 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 2 | 1

BASELINE CHARACTERISTICS:
Population: All participants who received at least one dose of study drug. Per protocol and statistical analysis plan (SAP), the primary and secondary analysis were performed to compare all tadalafil participants together versus all placebo participants together.
Groups:
- Tadalafil: Period 1: 20 mg middle weight cohort or 40 mg for heavy weight cohort administered orally by tablets once a day.
- Total: Total of all reporting groups
Arm/Group | Placebo | Tadalafil | Total
Number analyzed (Participants) | 18 | 17 | 35
Age, Continuous [Mean (Standard Deviation); unit: years] | 12.8 (3.39) | 14.1 (3.49) | 13.5 (3.45)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 10 | 19
  Male | 9 | 7 | 16
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7 | 8 | 15
  Not Hispanic or Latino | 6 | 4 | 10
  Unknown or Not Reported | 5 | 5 | 10
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 3 | 4
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 1 | 3
  White | 14 | 12 | 26
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Japan | 1 | 1 | 2
  Turkey | 2 | 1 | 3
  Brazil | 9 | 6 | 15
  Mexico | 1 | 4 | 5
  Israel | 2 | 4 | 6
  France | 1 | 1 | 2
  Germany | 1 | 0 | 1
  Poland | 1 | 0 | 1
6 Minute Walk Distance [Mean (Standard Deviation); unit: Meters] | 476.7 (105.11) | 485.8 (160.231) | 481.1 (132.77)

OUTCOME MEASURES:

1. Primary Outcome: Period 1: Change From Baseline to Week 24 in a 6 Minute Walk (MW) Distance in Meters
Description: 6MWD in meters assessed in a subset of participants who are ≥6 to <18 years of age who are developmentally capable of performing a 6MW test. Change from baseline was derived using mixed model repeated measures (MMRM) with terms for treatment group, visit, baseline 6MWD, and treatment-by-visit interaction.
Time Frame: Baseline, Week 24
Population: All participants who received at least one dose of study drug who were > = 6 to < 18 years of age and were capable of performing a 6MW test.
Measure: Least Squares Mean (Standard Error); unit: Meters
Arm/Group | Placebo | Tadalafil
Number analyzed (Participants) | 15 | 15
Meters | 36.60 (20.776) | 60.48 (20.410)
Statistical Analysis 1: Comparison: Placebo vs Tadalafil; Test type: Superiority; Mean Difference (Final Values) = 23.88, 80% CI 2-sided [-14.25 to 62.00], Standard Error of Mean 29.114

2. Secondary Outcome: Period 1: Time to Adjudicated Clinical Worsening (CW)
Description: Clinical worsening was defined as any of the following: death,lung or heart transplantation,atrial septostomy or Potts' shunt,hospitalization for Pulmonary Arterial Hypertension(PAH) progression,new onset syncope,initiation of new PAH therapy(including increase in the dose of existing PAH specific concomitant therapy,such as endothelin receptor agonist or beraprost medication), or increase of 1 or more in World Health Organization(WHO) Functional Class(except for participants already in Class IV;only for participants unable to perform the 6 minute walk(6MW) test;worsening of WHO functional class by 1 or more for participants who can perform a 6 minute walk(6MW) test and who have a decrease of ≥ 20% in the 6 minute walk distance(for those participants who are ≥6 years of age). Criteria for CW(from Period 1) were adjudicated by an independent,blinded study-specific Clinical Endpoint Committee(CEC).This adjudication was used for data analysis, and was not used to guide subject treatment.
Time Frame: Baseline through Week 24
Population: All participants who received at least one dose of study drug.
Measure: Median (95% Confidence Interval); unit: Weeks
Arm/Group | Placebo | Tadalafil
Number analyzed (Participants) | 18 | 17
Weeks | NA [NA to NA] — There was no confirmed adjudicated CW case to report. | NA [NA to NA] — There was no confirmed adjudicated CW case to report.

3. Secondary Outcome: Period 1: Percentage of Participants Who Experience CW
Description: Clinical worsening was defined as any of the following: death,lung or heart transplantation,atrial septostomy or Potts' shunt,hospitalization for Pulmonary Arterial Hypertension(PAH) progression,new onset syncope, initiation of new PAH therapy(including increase in the dose of existing PAH specific concomitant therapy,such as endothelin receptor agonist or beraprost medication),or increase of 1 or more in World Health Organization(WHO) Functional Class(except for participants already in Class IV; only for participants unable to perform the 6 minute walk(6MW) test;worsening of WHO functional class by 1 or more for participants who can perform a 6 minute walk(6MW) test and who have a decrease of ≥ 20% in the 6 minute walk distance(for those participants who are ≥6 years of age).Criteria for CW(from Period 1) were adjudicated by an independent,blinded study-specific Clinical Endpoint Committee(CEC).This adjudication was used for data analysis, and was not used to guide subject treatment.
Time Frame: Baseline through Week 24
Population: All participants who received at least one dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Tadalafil
Number analyzed (Participants) | 18 | 17
percentage of participants | 0 | 0

4. Secondary Outcome: Period 1: Pharmacokinetics (PK): Apparent Clearance (CL/F) of Tadalafil at Steady-state
Description: Period 1: Pharmacokinetics (PK): Apparent Clearance (CL/F) of Tadalafil at steady-state
Time Frame: Week 2, Week 4, Week 16 and Week 24
Population: All participants who received at least one dose of study drug and had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liter Per Hour (L/hr)
Groups:
- 20 mg Tadalafil: Period 1: 20 mg tadalafil administered orally by tablets once a day with concomitant endothelin receptor antagonist (ERA).
- 40 mg Tadalafil: Period 1: 40 mg tadalafil administered orally by tablets once a day with concomitant ERA.
Arm/Group | 20 mg Tadalafil | 40 mg Tadalafil
Number analyzed (Participants) | 4 | 13
Liter Per Hour (L/hr)
  With concomitant bosentan: number analyzed (Participants) | 3 | 13
  With concomitant bosentan | 3.63 (38.1) | 4.49 (28.2)
  No bosentan (ERA: Macitentan): number analyzed (Participants) | 1 | 0
  No bosentan (ERA: Macitentan) | NA (NA) — For n = 1, geometric mean and geometric coefficient of variation could not be calculated. Individual value is 2.68. |

5. Secondary Outcome: Period 2: Percentage of Participants Who Experience CW
Description: Clinical worsening was defined as any of the following: death, lung or heart transplantation, atrial septostomy or Potts' shunt, hospitalization for Pulmonary Arterial Hypertension (PAH) progression, new onset syncope, initiation of new PAH therapy (including increase in the dose of existing PAH specific concomitant therapy, such as endothelin receptor agonist or beraprost medication), or increase of 1 or more in World Health Organization(WHO) Functional Class (except for participants already in Class IV; only for participants unable to perform the 6 minute walk (6MW) test; worsening of WHO functional class by 1 or more for participants who can perform a 6 minute walk (6MW) test and who have a decrease of ≥ 20% in the 6 minute walk distance (for those participants who are ≥6 years of age).
Time Frame: Period 2 Baseline through Study Completion (Up to 24 Months)
Population: Period 2: All participants who received at least one dose of study drug.
Measure: Number; unit: percentage of participants
Groups:
- Placebo/Tadalafil - Open-Label Treatment: Period 2: 20 mg middle weight cohort or 40 mg for heavy weight cohort administered tadalafil orally by tablets once a day.
  Participants had received placebo during period 1.
- Tadalafil/Tadalafil - Open-Label Treatment: Period 2: 20 mg middle weight cohort or 40 mg for heavy weight cohort administered tadalafil orally by tablets once a day.
  Participants had received tadalafil during period 1.
Arm/Group | Placebo/Tadalafil - Open-Label Treatment | Tadalafil/Tadalafil - Open-Label Treatment
Number analyzed (Participants) | 16 | 16
percentage of participants | 12.5 | 18.8

6. Secondary Outcome: Period 2: Time to First Occurrence of CW
Description: as for outcome 5
Time Frame: Period 2 Baseline through Study Completion (Up to 24 Months)
Population: Period 2: All participants who received at least one dose of study drug, who entered the open-label treatment Period
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Placebo/Tadalafil - Open-Label Treatment | Tadalafil/Tadalafil - Open-Label Treatment
Number analyzed (Participants) | 16 | 16
Months | NA [NA to NA] — Median and CI are not estimable due to inadequate events of Clinical Worsening (CW) using Kaplan-Meier survival Estimates. | NA [NA to NA] — Median and CI are not estimable due to inadequate events of Clinical Worsening (CW) using Kaplan-Meier survival Estimates.

ADVERSE EVENTS:
Time Frame: Baseline Up To 24 Months
Description: All participants who received at least one dose of study drug. Gender specific events only occurring in male or female participants have had the number of participants at risk adjusted accordingly.
Groups:
- Placebo - Double Blind: Period 1: Participants received placebo orally by tablets once a day.
- Tadalafil - Double Blind: Period 1: 20 mg middle weight cohort or 40 mg for heavy weight cohort administered tadalafil orally by tablets once a day.
Arm/Group | Placebo - Double Blind | Tadalafil - Double Blind | Placebo/Tadalafil - Open-Label Treatment | Tadalafil/Tadalafil - Open-Label Treatment
All-Cause Mortality (participants affected / at risk) | 0/18 | 0/17 | 0/16 | 0/16
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/17 | 4/16 | 1/16
Other Adverse Events (participants affected / at risk) | 8/18 | 15/17 | 11/16 | 12/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo - Double Blind (N=18) | Tadalafil - Double Blind (N=17) | Placebo/Tadalafil - Open-Label Treatment (N=16) | Tadalafil/Tadalafil - Open-Label Treatment (N=16)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Acute right ventricular failure (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Placebo - Double Blind (N=18) | Tadalafil - Double Blind (N=17) | Placebo/Tadalafil - Open-Label Treatment (N=16) | Tadalafil/Tadalafil - Open-Label Treatment (N=16)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Eosinophilia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Palpitations (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ventricular extrasystoles (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Asthenopia (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Photopsia (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Dental caries (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Enterocolitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Irritable bowel syndrome (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Plicated tongue (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Asthenia (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Exercise tolerance decreased (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypersensitivity (Immune system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Seasonal allergy (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Acute sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Ascariasis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Body tinea (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ear infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Impetigo (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 3 (3) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (2) | 3 (4)
Otitis media acute (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Paronychia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pharyngitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 2 (4)
Rhinitis (Infections and infestations) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Sinusitis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 1 (2)
Tonsillitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tracheobronchitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 3 (3) | 0 (0) | 2 (2)
Urinary tract infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Vaginal infection (Infections and infestations) | 0/9 (0) | 1/10 (1) | 0/8 (0) | 0/10 (0)
Viral infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Viral tonsillitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Viral upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bone contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Penis injury (Injury, poisoning and procedural complications) | 0/9 (0) | 0/7 (0) | 1/8 (1) | 0/6 (0)
Blood creatine phosphokinase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hepatic enzyme increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dyslipidaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vitamin b12 deficiency (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vitamin d deficiency (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2) | 0 (0) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Patellofemoral pain syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pharyngeal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 3 (3)
Headache (Nervous system disorders) | 2 (6) | 5 (5) | 2 (2) | 3 (3)
Presyncope (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Somnolence (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Excessive masturbation (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Menorrhagia (Reproductive system and breast disorders) | 0/9 (0) | 1/10 (1) | 1/8 (1) | 1/10 (2)
Metrorrhagia (Reproductive system and breast disorders) | 0/9 (0) | 0/10 (0) | 0/8 (0) | 1/10 (1)
Penis disorder (Reproductive system and breast disorders) | 0/9 (0) | 1/7 (1) | 0/8 (0) | 0/6 (0)
Polymenorrhoea (Reproductive system and breast disorders) | 0/9 (0) | 0/10 (0) | 0/8 (0) | 1/10 (1)
Spontaneous penile erection (Reproductive system and breast disorders) | 0/9 (0) | 1/7 (2) | 1/8 (1) | 0/6 (0)
Uterine haemorrhage (Reproductive system and breast disorders) | 0/9 (0) | 0/10 (0) | 1/8 (1) | 0/10 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 1 (1) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Pulmonary arterial hypertension (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Haemorrhage subcutaneous (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (3) | 0 (0) | 0 (0)
Livedo reticularis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Swelling face (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Menarche (Social circumstances) | 1/9 (1) | 0/10 (0) | 0/8 (0) | 0/10 (0)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Flushing (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
The study is mainly descriptive in a small number of children with PAH and there were no participants enrolled in the light weight cohort.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2018-12-13): https://cdn.clinicaltrials.gov/large-docs/90/NCT01824290/Prot_000.pdf
  • Statistical Analysis Plan (2019-03-28): https://cdn.clinicaltrials.gov/large-docs/90/NCT01824290/SAP_001.pdf